CLINICAL TRIAL: NCT01986673
Title: Single-Dose Relative Bioavailability Study of SST-6006, a Topical Sildenafil Cream Versus Oral Sildenafil in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SST-6006-001-01
Record Dates: First submitted 2013-10-29; First posted 2013-11-18 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Pharmacokinetic Characterization
MeSH Terms: interventions — Sildenafil Citrate

ARMS (2):
- 5% Sildenafil Cream (SST-6006) (Experimental): 5% Sildenafil Cream
  Interventions: Drug: 5% Sildenafil Cream (SST-6006)
- Oral Sildenafil 50 mg (Active Comparator): Oral Sildenafil 50 mg
  Interventions: Drug: Oral Sildenafil 50 mg

INTERVENTIONS:
Drug: 5% Sildenafil Cream (SST-6006) — 5 % Sildenafil Cream
  Arms: 5% Sildenafil Cream (SST-6006)
Drug: Oral Sildenafil 50 mg — Oral Sildenafil 50 mg
  Arms: Oral Sildenafil 50 mg

SUMMARY:
The purpose of this study is to evaluate how a single dose of sildenafil cream (SST-6006) is absorbed and eliminated by the body, with and without the use of a condom, compared to a single oral sildenafil dose and to evaluate the safety of sildenafil cream.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign and date the written informed consent form (ICF) before any study-specific screening procedures are performed
2. Men between the ages of 18 to 55 years, inclusive
3. Body mass index (BMI = weight [kg]/height [m]2) between 18.0 to 30.0 kg/m2, inclusive and body weight of at least 50 kg
4. Nonsmoker or past smoker who has been abstinent for 6 months before study Day 1
5. Have a high probability for compliance with and completion of the study, in the opinion of the Principal Investigator
6. Healthy as determined by the investigator based on medical history, physical examination, clinical laboratory tests, vital sign measurements, and a normal 12-lead ECG
7. Resting supine systolic blood pressure between 90 and 140 mmHg and resting supine diastolic blood pressure between 50 and 90 mmHg
8. Must be able to achieve a successful erection

Exclusion Criteria:

1. Presence or history of any disorder that may prevent the successful completion of the study
2. Presence of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or psychiatric disease, or other unstable medical condition
3. Subjects with a history of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to study Day 1, or a history of coronary disease causing angina
4. Subjects with retinitis pigmentosa and subjects with sickle cell anemia or related anemias, even if they feel clinically well at the time of screening. Subjects with retinitis pigmentosa will be identified by specifically asking whether they have the condition, if there are visual signs and symptoms of the condition (including questioning subjects as to whether they have difficulty seeing at night or in low light, and if they have any visual field deficits that indicate a loss of peripheral or central vision), or if there is a family history
5. Subjects with anatomical deformations of the penis such as angulation, cavernosal fibrosis or Peyronie's disease
6. History of orthostatic hypotension or orthostatic hypotension present at the screening visit, defined as a drop in systolic blood pressure greater than 20 mm Hg and a drop in diastolic blood pressure greater than 10 mm Hg with a change in position from supine to standing
7. A history of erectile dysfunction or a prostatectomy
8. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article
9. Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study Day 1
10. History of drug abuse within 1 year before study Day 1
11. History of alcoholism within 1 year before study Day 1, admitted alcohol abuse, or average consumption of more than 2 standard units of alcohol per day (a standard unit equals 12 ounces of beer, 1½ ounces of 80-proof alcohol, or 6 ounces of wine)
12. Use of any prescription drugs within 28 days before study Day 1, or over-the-counter drugs, including herbal supplements (except for the occasional use of acetaminophen [Tylenol] and vitamins) within 14 days before study Day 1. If the subject takes any prescription or OTC drugs at the direction of a health care provider, that provider should be consulted before medications are stopped for the purposes of study participation.
13. Positive serologic findings for human immunodeficiency virus antibodies (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HCV)
14. Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, and opiates) or alcohol screen
15. Participation in a clinical trial within 30 days before study Day 1
16. Consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours before study Day 1
17. Consumption of grapefruit or grapefruit-containing products within 72 hours before study Day 1
18. Any skin breaks, irritation, or lesions present in the area to which the cream will be applied, assessed at screening and check-in
19. A drug or food allergy which in the opinion of the Investigator contraindicates participation in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, AUC 0-tlast, AUC 0-t, Kel, AUC0-inf, t1/2, CL/F | 32 hours

SECONDARY OUTCOMES:
Adverse Events | 7 to 10 days
  Number of subjects experiencing TEAEs.
Clinical Chemistry Tests | 1 day
  Changes from baseline in clinical chemistry values
Vital Signs | 1 day
  Vital sign changes from pre-dose

CONTACTS AND LOCATIONS:
Locations (1):
- SST Clinical Site, Miami, Florida, United States